CLINICAL TRIAL: NCT07055464
Title: Comparative Study Between Etep-rs and Ipom Plus for Abdominal Wall Hernias
Brief Title: Comparison Between eTEP-RS vs IPOM PLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GSVM Medical College (Other)
Responsible Party: Principal Investigator, Kavita Sijwali, Junior resident, DEPARTMENT OF GENERAL SURGERY, GSVM Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETEPIPOM2024
Record Dates: First submitted 2025-06-19; First posted 2025-07-09 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Ventral Hernia Repair; Abdominal Hernia
Keywords: Etep-rs and ipom plus; Ventral hernia; Mesh repair
MeSH Terms: conditions — Hernia, Abdominal; Hernia, Ventral | interventions — Herniorrhaphy

STUDY DESIGN:
Intervention Model Description: Two-arm parallel group randomized controlled trial comparing eTEP-RS and IPOM Plus for elective abdominal wall hernia repair. Eligible participants are randomly assigned to one of the two surgical techniques. Both groups are followed in parallel to assess intraoperative, postoperative, and follow-up outcomes including pain, hospital stay, complications, and recurrence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eTEP-RS Technique (Experimental): Patients undergoing laparoscopic abdominal wall hernia repair using the eTEP-RS (Enhanced View Totally Extraperitoneal-Retromuscular) technique.
  Interventions: Procedure: eTEP-RS Hernia Repair
- IPOM Plus Technique (Active Comparator): Patients undergoing laparoscopic abdominal wall hernia repair using the IPOM Plus technique with fascial defect closure.
  Interventions: Procedure: IPOM Plus Hernia Repair

INTERVENTIONS:
Procedure: eTEP-RS Hernia Repair — Laparoscopic retromuscular mesh repair using the enhanced view totally extraperitoneal (eTEP-RS) technique for ventral or incisional hernia.
  Arms: eTEP-RS Technique
Procedure: IPOM Plus Hernia Repair — Intraperitoneal onlay mesh (IPOM Plus) repair involving laparoscopic fascial defect closure and mesh placement for abdominal wall hernias.
  Arms: IPOM Plus Technique

SUMMARY:
This study aims to compare the outcomes of Enhanced View Totally Extraperitoneal Rives-Stoppa (eTEP-RS) repair and Intraperitoneal Onlay Mesh Plus (IPOM Plus) repair in the management of ventral wall hernias. The comparison includes operative time, post-operative pain, hospital stay, surgical site occurrences, and recurrence rates. Patients will be prospectively enrolled and allocated into two groups based on the surgeon's discretion or patient-specific criteria.

DETAILED DESCRIPTION:
Abdominal wall hernias are common surgical conditions, and multiple techniques have evolved for their repair. eTEP-RS is a relatively newer, minimally invasive approach that combines the principles of the Rives-Stoppa retromuscular mesh placement with the benefits of laparoscopic surgery. IPOM Plus, on the other hand, is a widely practiced technique involving intraperitoneal mesh placement with defect closure.

This prospective comparative study is designed to evaluate the effectiveness and safety of eTEP-RS versus IPOM Plus in patients undergoing elective repair of ventral or incisional hernias. The study will assess intra-operative parameters (e.g., duration of surgery, blood loss), early post-operative outcomes (pain score, duration of hospital stay), surgical site complications (seroma, infection, mesh-related issues), and long-term outcomes (recurrence, quality of life).

Patients fulfilling inclusion criteria will be assigned to one of the two arms. Standardized protocols will be followed for pre-operative work-up, anesthesia, surgical steps, and post-operative care. Data will be analyzed to determine if one technique offers superior clinical outcomes, better patient satisfaction, or reduced recurrence

ELIGIBILITY:
Inclusion Criteria:

* patient with uncomplicated ventral hernia with defect size between 2 cm and 5 cm
* Age between 18 years and 60 years.
* elective surgical cases(non emergency)

Exclusion Criteria:

* defect size greater than 5 cm.
* patient not giving consent.
* patient with lateral HERNIAS.
* patient with complicated ventral HERNIAS like irreducible , obstructed and strangulated HERNIAS.
* pregnant and lactating women.
* patient on anticoagulants.
* recurrent hernia.
* patient not fit for GA.
* POOR GENERAL CONDITION.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Hernia Recurrence Rate | Up to 6 months post-surgery
  Clinical or radiological evidence of hernia recurrence during follow-up.
Postoperative Pain Score | 6 months
  Postoperative pain will be assessed using the Visual Analogue Scale (VAS) 24 hours, and 7 days, 30 days and 6 months after surgery.
  Pain intensity will be assessed using the Visual Analog Scale (VAS). The scale ranges from 0 to 10, where:
  0 = No pain
  10 = Worst imaginable pain Higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Operative Time | Intraoperative
  Time from first incision to final closure, measured in minutes.
Duration of Postoperative Hospital Stay | DAY 1 TO DAY 15
  Number of days from surgery to discharge(upto 15 days post- operatively)
Incidence of Surgical Site Occurrences (SSOs) | Within 30 days post-surgery
  Includes wound infection, seroma, hematoma, or mesh-related complications occurring within 30 days
Time to Return to Normal Activities | Within 30 days postoperatively
  Number of days taken by the patient to resume routine daily activities, such as walking without support, household tasks, or returning to work, as reported during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Sijwali, MBBS, MS SURGERY RESIDENT, Principal Investigator — GSVM MEDICAL COLLEGE KANPUR
Locations (1):
- Gsvm Medical College Kanpur, Kanpur, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
The Inpatient Department (IPD) of the Department of General Surgery is used by multiple researchers. However, patients eligible for this study will be screened using a separate screening log. Only patients meeting the inclusion criteria and providing informed written consent will be enrolled. No overlap in participant enrollment with other interventional trials will occur. Ethical clearance has been obtained and institutional guidelines for shared clinical spaces will be followed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after primary study completion date to 5 years after study completion
Access Criteria: Qualified researchers, academicians, and clinicians may request access to de-identified individual participant data (IPD) and supporting information including the study protocol, informed consent form (ICF), and statistical analysis plan (SAP) after the primary results have been published.
  Access will be provided upon reasonable request submitted via email to the Principal Investigator. Requests must include a summary of the intended use and a data-sharing agreement to ensure compliance with confidentiality and ethical standards.
  No personally identifiable data will be shared. The information will be made available through secure institutional email correspondence or a protected data-sharing platform, subject to Institutional Ethics Committee approval if required.
URL: https://notapplicable.example.com

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT07055464/Prot_SAP_000.pdf